CLINICAL TRIAL: NCT05632419
Title: Assess the 6-month Prognosis of Patients Who Presented With a State of Extreme Agitation: "Excited Delirium Syndrome" AGICOHORT
Brief Title: Prognosis of Patients Who Presented With a State of Extreme Agitation.
Acronym: AGICOHORT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Lariboisière-Saint Louis clinical research unit (Unknown)
Responsible Party: Sponsor
Other Study IDs: P220382
Record Dates: First submitted 2022-10-28; First posted 2022-11-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to assess the 6-month prognosis of patients who presented with extreme agitation in the emergency room.

The primary endpoint is the 6-month mortality of agitated patients.

DETAILED DESCRIPTION:
Emergency services are confronted with emergency situations characterized by patients who are victims of significant agitation, in particular states of extreme agitation "excited delirium syndrome", which is constantly increasing and which seems to be associated with morbidity and mortality not negligible.

Patients meeting the inclusion and non-inclusion criteria are included on admission to the emergency room.

An evaluation at H1 and at the end of hospitalization is carried out. The patient is contacted by telephone at M1, M3 and M6.

The inclusion period is 24 months The duration of participation (treatment + follow-up) is 6 months The total duration is 30 months.

The research is multicentric and national with the participation of 8 centres.

ELIGIBILITY:
Inclusion Criteria:

* Agitated patient with the presence of three major criteria, namely,
* restlessness
* insensitivity to pain
* tachypnea (fr>20)

and the presence of a minor criterion among

* sweating
* skin hyperthermia
* non-compliance with law enforcement
* tirelessness
* unusual strength
* inappropriate clothing, nudity

Exclusion Criteria:

* patient age < 18 years
* head trauma
* pregnancy
* detained
* other obvious causes of pain leading to restlessness (renal colic, migraines, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Agitated patients
Sampling Method: Probability Sample
Enrollment: 608 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2027-01-17 (Estimated); Study Completion 2027-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of deceased patients | 6 months
  The 6-month prognosis of patients who presented with extreme agitation in the emergency room.

SECONDARY OUTCOMES:
Assess the characteristics of agitated patients regarding the age | 6 months
  Age
Assess the characteristics of agitated patients regarding the gender | 6 months
  Gender
Assess the characteristics of agitated patients regarding the mode of arrival in the emergency room | 6 months
  Mode of arrival in the emergency room
Assess the characteristics of agitated patients regarding medical history | 6 months
  Medical history
Assess the characteristics of agitated patients regarding vital signs (blood pressure) | 6 months
  Blood pressure
Assess the characteristics of agitated patients regarding vital signs (oxygen saturation) | 6 months
  Oxygen saturation
Assess the characteristics of agitated patients regarding vital signs (heart rate) | 6 months
  Heart rate
Assess the characteristics of agitated patients regarding vital signs (respiratory rate) | 6 months
  Respiratory rate
Assess the characteristics of agitated patients regarding vital signs (temperature) | 6 months
  Temperature
Assess the characteristics of agitated patients regarding vital signs (Glasgow coma scale) | 6 months
  Glasgow coma scale (The GCS is scored between 3 and 15, 3 being the worst and 15 the best).
Assess the characteristics of agitated patients regarding vital signs (Corrected QT interval on electrocardiogram) | 6 months
  Corrected QT interval (QTc)
Assess the characteristics of agitated patients regarding patient biology (blood ionogram) | 6 months
  Blood ionogram
Assess the characteristics of agitated patients regarding patient biology (urine and blood toxins) | 6 months
  Urine and blood toxins
Assess the characteristics of agitated patients regarding patient biology | 6 months
  Arterial blood gas
Assess the characteristics of agitated patients regarding patient biology (Complete blood count) | 6 months
  Complete blood count (CBC)
Assess the characteristics of agitated patients regarding agitation (RASS) | 6 months
  Agitation assessment scale (Richmond Agitation Sedation Scale, RASS) (-5 = worse outcome to +4 = worse outcome, 0 is the better outcome)
Assess the characteristics of agitated patients regarding agitation (BARS) | 6 months
  Agitation assessment scale (Behavioural Activity Rating Scale, BARS) (1 = worse outcome to 7 = worse outcome , 4 is the better outcome)
Assess the characteristics of agitated patients regarding agitation (CGI S) | 6 months
  Agitation assessment scale (Clinical Global Impression Severity or CGI S, 0 = Not evaluated to 7 = worse outcome)
Characterize the etiologies of this syndrome (organic, psychiatric or iatrogenic) | 6 months
  Organic
  * medical background,
  * somatic etiology research with intrinsic imputability criteria (chronological and semiological) and extrinsic (literature)
  * capillary blood glucose, temperature, Glasgow, electrocardiogram
  * blood ionogram, arterial blood gas, blood count Iatrogenic
  * analytical by means of a urinary and blood toxin screening for recent consumptions of psychoactive substances
  * search the treatment of the patient psychiatric
  * clinical observations obtained during consultation
Characterize the management of patients in extreme agitation according to initial pharmacological treatments administered | 6 months
  Initial pharmacological treatments administered
Characterize the management of patients in extreme agitation according to the need for physical restraints | 6 months
  Need for physical restraints
Characterize the management of patients in extreme agitation according to the eed for upper airway protection with intubation | 6 months
  Need for upper airway protection with intubation
Assess the efficacy of the pharmacological treatments administered (GCI S) | 6 months
  According to agitation scale at H1, H2 (Clinical Global Impression Severity or CGI S, 0 = Not evaluated to 7 = worse outcome) and need for other pharmacological treatments
Assess the efficacy of the non-pharmacological treatments administered (RASS) | 6 months
  According to agitation scale at H1, H2 (Richmond Agitation Sedation Scale, RASS) (-5 = worse outcome to +4 = worse outcome, 0 is the better outcome) and need for other non-pharmacological treatments
Assess the efficacy of the non-pharmacological treatments administered (BARS) | 6 months
  According to agitation scale at H1, H2 (Behavioural Activity Rating Scale, BARS) (1 = worse outcome to 7 = worse outcome , 4 is the better outcome) and need for other non-pharmacological treatments

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Adnet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Avicenne Hospital - Aphp, Bobigny, Île-de-France Region, France